CLINICAL TRIAL: NCT06132594
Title: Computed Guided Prolotherapy Versus Conventional Prolotherapy in Treatment of TMJ Internal Derangment
Brief Title: Computed Guided Prolotherapy Versus Conventional Prolotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Zahran Arafat Ahmed Arafat, Demonstrator at the Department of oral and Maxillofacial Surgery, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUAREC20210100-09
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Temporomandibular Joint Disorders; Orofacial Pain
Keywords: TMD; Temporomandibular Joint Disorders; Prolotherapy of TMJ; Guided Arthrocentesis
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I; Conventional arthrocentesis followed by I-PRF injection (Experimental): Patients received arthrocentesis followed by I-PRF injection, employing the conventional TMJ injection technique aided by facial anatomical landmarks
  Interventions: Procedure: Conventional arthrocentesis followed by I-PRF injection
- Group II; 3d surgical guided Arthrocentesis followed by I-PRF injection (Experimental): Patients received arthrocentesis followed by I-PRF injection with the assistance of a CT-guided 3D printed surgical guide.
  Interventions: Procedure: 3d surgical guided Arthrocentesis followed by I-PRF injection

INTERVENTIONS:
Procedure: Conventional arthrocentesis followed by I-PRF injection — An auriculotemporal nerve block using Mebacaine 0.5% was administered near the mandible's neck. The patient sat at a 45° angle with their head turned. The posterior entry point was 10 mm from the midtragus and 2 mm below the line, while the anterior entry point was marked 20 mm from the midtragus and 10 mm below the line. A biting block kept the mouth open. 2-3 ml of Ringer lactate was injected with an 18-gauge needle to enlarge the joint space. A second needle allowed the solution to flow freely. After lavaging the joint, 1 ml of I-PRF was injected into the upper joint space. Jaw manipulation was done to address adhesions and improve disc mobility.
  Arms: Group I; Conventional arthrocentesis followed by I-PRF injection
Procedure: 3d surgical guided Arthrocentesis followed by I-PRF injection — Patients underwent arthrocentesis with Ringer lactate, followed by I-PRF injection in the TMJ's superior space using a CT-planned 3D-printed guide. Positioned at a 45° angle, patients were comfortably seated, and disinfection was performed. The patient-specific guide, fitting over maxillary teeth and the face, was employed unilaterally or bilaterally with a biting block for mouth opening maintenance. An 18-gauge needle administered 2-3 ml of Ringer lactate, widening the joint space, followed by a second needle allowing free solution flow (80-90 ml) to flush the superior joint space. Post-arthrocentesis, 1 ml of I-PRF was injected. To enhance joint mobility and free the disc, gentle manipulation of the lower jaw was performed after removing the needles and guide.
  Arms: Group II; 3d surgical guided Arthrocentesis followed by I-PRF injection

SUMMARY:
The aim of that study is to compare between conventional prolotherapy and computed guided prolotherapy in treatment of temporomandibular joint (TMJ) internal derangement.

DETAILED DESCRIPTION:
This study will include patients with TMJ internal derangement with signs and symptoms of pain, clicking and limited mouth opening .The study will be held in oral and maxillofacial department, Faculty of Dental Medicine, Al-Azhar University, Assiut branch. Internal derangement of the joint will be confirmed by magnetic resonance image (MRI).

Patients included in this study will be divided randomly into two equal groups by the aid of financial coins. Group I: patients will be conventionally injected into the superior space of TMJ by injectable PRF by the aid of the surface facial landmarks where the patient will seated comfortably at 45° angle on the dental chair with the head turned toward the unaffected side. The target site will be prepared and disinfected with betadine. The points of needle insertion will be marked on the skin according to a line will be draw from the middle of the tragus of the ear to the outer canthus of the eye and entry points will be marked along this cantho-tragal line which will correspond to the glenoid fossa and will be marked 10 mm from the mid-tragus and 2 mm below the line.

Group II: patients will be injected into the superior space of TMJ with I- PRF by the aid of specific CT-planned 3D-printed surgical guide, which will lead the needle insertion, and the accuracy of the needle insertion into the superior space of the TMJ will be assessed.

Preparation of I-PRF:

The cubital area of the patient arm will be disinfected with betadine and the blood will be drawn from the patient cubital vein into plain tubes (vaccutainers) under aseptic conditions .The loaded tubes will be centrifuged at 750 rpm for 3 minutes and the I-PRF will be aspirated into a plastic syringe to be ready for injection into the superior space of the TMJ of patients of each group.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral or unilateral TMJ internal derangement.
* No response to conservative treatments (soft diet, occlusal splint, muscle relaxants, non-steroidal anti-inflammatory drugs, or movement restriction).
* Ability to undergo MRI or CT scans without contraindications.

Exclusion Criteria:

* Those with systemic diseases (polyarthritis or rheumatoid diseases).
* Individuals with neurologic disorders.
* Patients with a history of condylar fracture or previous TMJ injections.
* Those with head and neck cancer.
* Completely edentulous patients (lacking teeth).
* Individuals with implanted metal or medical devices.
* Patients with developmental and congenital disorders of the TMJ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain | Intraoperative,1 week, 1month and 3 months
  Using visual analog scale
The number of needle insertion attempts | Intraoperative
  The number of needle insertions, indicative of the attempts, was counted for each group.

SECONDARY OUTCOMES:
Maximal incisal opening | 1 week, 1month and 3 months
  Using digital caliper in Millimeter (mm)
Time of operation | Intraoperative
  In minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine - Al-Azhar University, Asyut, Egypt

REFERENCES:
- [Background] Young AL. Internal derangements of the temporomandibular joint: A review of the anatomy, diagnosis, and management. J Indian Prosthodont Soc. 2015 Jan-Mar;15(1):2-7. doi: 10.4103/0972-4052.156998. PMID 26929478
- [Background] Laskin DM. Arthroscopy Versus Arthrocentesis for Treating Internal Derangements of the Temporomandibular Joint. Oral Maxillofac Surg Clin North Am. 2018 Aug;30(3):325-328. doi: 10.1016/j.coms.2018.04.008. Epub 2018 Jun 1. PMID 29866452
- [Background] Custodio ALN, Cameron A, Bakr M, Little C, Chrcanovic BR, Reher P. Positioning accuracy assessment of minimally invasive percutaneous injection techniques for the treatment of temporomandibular disorders. Dentomaxillofac Radiol. 2021 Feb 1;50(2):20200313. doi: 10.1259/dmfr.20200313. Epub 2020 Jul 24. PMID 32706994
- [Background] Sivri MB, Ozkan Y, Pekiner FN, Gocmen G. Comparison of ultrasound-guided and conventional arthrocentesis of the temporomandibular joint. Br J Oral Maxillofac Surg. 2016 Jul;54(6):677-81. doi: 10.1016/j.bjoms.2016.04.004. Epub 2016 Apr 23. PMID 27118616
- [Background] Mahmoud K, Galal N, Ali S, Gibaly A, Elbehairy MS, Mounir M. Computer-Guided Arthrocentesis Using Patient-Specific Guides: A Novel Protocol for Treatment of Internal Derangement of the Temporomandibular Joint. J Oral Maxillofac Surg. 2020 Mar;78(3):372.e1-372.e7. doi: 10.1016/j.joms.2019.10.005. Epub 2019 Oct 15. PMID 31705867
- [Background] Hyder A, Tawfik BE, Elmohandes W. Efficacy of computer-guided versus conventional sodium hyaluronate injection in superior joint space in treatment of temporomandibular joint (TMJ) internal derangement: Comparative randomized controlled trial. J Stomatol Oral Maxillofac Surg. 2022 Oct;123(5):e321-e326. doi: 10.1016/j.jormas.2022.05.007. Epub 2022 May 8. PMID 35545190